CLINICAL TRIAL: NCT04259307
Title: Effect of Intensive Nutritional Support on Functional Recovery in Subacute Stroke Patient
Brief Title: Effect of Intensive Nutritional Support in Subacute Stroke Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Korean Center for Disease Control and Prevention (Other Government)
Responsible Party: Principal Investigator, Won Hyuk Chang, Associate Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-06-109
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Stroke; Rehabilitation; Nutrition
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive nutrition group (Experimental): Standard nutritional support with additional intravenous nutrition of 500 kcal per day for 3 weeks
  Interventions: Drug: Omapone Peri 724mL or Winuf Peri 654mL
- Control group (No Intervention): Standard nutritional support only per day for 3 weeks

INTERVENTIONS:
Drug: Omapone Peri 724mL or Winuf Peri 654mL — Additional intravenous nutrition of 500 kcal per day for 3 weeks
  Other Names: Comprehensive rehabilitation
  Arms: Intensive nutrition group

SUMMARY:
Proper nutritional support during early rehabilitation may be beneficial for functional improvements in gaining functional independence and preventing complications in stroke patients. However, there was no consensus of proper amount of nutritional support in stroke patients. In this study, the investigators aimed to clarigy the effects of the intensive nutritional support during comprehensive rehabilitation during subacute phase to improve function in patients with first-ever strokes.

ELIGIBILITY:
Inclusion Criteria:

* Acute first-ever stroke patients less than 7 days after onset

  * more than 19 years old at stroke onset ③ stroke confirmed by brain CT or MRI

    * body mass index (BMI) <25 before the comprehensive rehabilitation ⑤ Mini Nutritional Assessment < 12 before the comprehensive rehabilitation ⑥ Fugl-Meyer assessment < 85 at 7 days after stroke onset

Exclusion Criteria:

* Transient ischemic stroke

  * Progressive or unstable stroke

    * Pre-existing and active major neurological disease, e.g., spinal cord injury, Parkinson's disease, et al.

      * Pre-existing and active (e.g., on chronic medication) major psychiatric disease, such as major depression, schizophrenia, bipolar disease or dementia ⑤ Advanced liver, kidney, cardiac, or pulmonary disease, e.g., advanced hepatocellular carcinoma, end-stage renal failure, et al.)

        * A terminal medical diagnosis consistent with survival < 1 year

          * Diabetes mellitus, Hyperlipidemia, Metabolic syndrome, Heart failure) ⑧ Pregnant or lactating women ⑨ Prohibited from taking medication (Omapone Peri 724mL or Winuf Peri 654mL)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2020-01-29 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Korean modified Barthel Index (K-MBI) at 6 months after onset | 6 months after onset
  Korean modified Barthel Index (0~100)

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim DH, Sohn MK, Lee J, Kim DY, Shin YI, Oh GJ, Lee YS, Joo MC, Lee SY, Song MK, Han J, Ahn J, Lee HS, Kim YT, Kim YH, Chang WH. Effect of intensive nutritional support on functional recovery in subacute stroke: A randomized, multicenter, single-blinded trial. Ann Phys Rehabil Med. 2025 May;68(4):101976. doi: 10.1016/j.rehab.2025.101976. Epub 2025 Apr 17. PMID 40250062